CLINICAL TRIAL: NCT01057407
Title: A Phase 3, Multicenter, Open-label, Sevelamer Hydrochloride-controlled Study in Chronic Kidney Disease (CKD) Patients With Hyperphosphatemia on Hemodialysis
Brief Title: A Comparative Study of ASP1585 in Chronic Kidney Disease Patients With Hyperphosphatemia on Hemodialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1585-CL-0003
Record Dates: First submitted 2010-01-25; First posted 2010-01-27 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-04

CONDITIONS: Chronic Kidney Disease; Renal Dialysis; Renal Insufficiency
Keywords: Hyperphosphatemia; hemodialysis; CKD; ASP1585
MeSH Terms: conditions — Renal Insufficiency, Chronic; Renal Insufficiency; Hyperphosphatemia | interventions — Sevelamer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ASP group (Experimental)
  Interventions: Drug: ASP1585
- Sevelamer group (Active Comparator)
  Interventions: Drug: Sevelamer hydrochloride

INTERVENTIONS:
Drug: ASP1585 — oral
  Other Names: ILY101; AMG223
  Arms: ASP group
Drug: Sevelamer hydrochloride — oral
  Other Names: Renagel; phosbloc
  Arms: Sevelamer group

SUMMARY:
This is a multi-center, open-labeled study to examine the non-inferiority of ASP1585 to sevelamer hydrochloride in chronic kidney disease patients with hyperphosphatemia on hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney disease patients on hemodialysis
* Hyperphosphatemia
* Patients on a phosphate binder or phosphate lowering drug for 28 days or longer, and that, those for whom the dose has not been changed within 28 days
* Written informed consent

Exclusion Criteria:

* Patients with gastrointestinal surgery or enterectomy
* Patients with severe cardiac diseases
* Patients with severe constipation or diarrhea
* Patients with a history or complication of malignant tumors
* Patients with uncontrolled hypertension
* Patients treated with parathyroid intervention

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2010-01; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Serum phosphorus level at the end of treatment | After 12-week or at the treatment discontinuation

SECONDARY OUTCOMES:
Change in serum phosphorus level | After 12-week or at the end of treatment
Time-course changes in serum phosphorus levels | During Treatment
Changes in serum Ca x P | During treatment
Changes in intact PTH levels | During Treatment

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (3):
- Japan (3):
  - Chūbu
  - Kantou
  - Kyusyu

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086